CLINICAL TRIAL: NCT00577928
Title: Correlation of Fecal Calprotectin Level With the Clinical, Endoscopic, Histologic and Radiologic Activity in Inflammatory Bowel diseaseThe Value of Fecal Calprotectin for the Diagnosis and Assessment of Inflammatory Bowel Disease
Brief Title: Value of Fecal Calprotectin
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: 060362; IRB# 0603-62
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Calprotectin; Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
For the main goal - the accuracy of calprotectin for the diagnosis of IBD - calprotectin levels will be compared between patients with and without a diagnosis of IBD and the sensitivity, specificity and accuracy will be determined. For the secondary aim - the correlation between calprotectin levels and disease activity - in patients with IBD selected from this cohort, we will determine the association between calprotectin levels and clinical IBD score, serological markers (WBC, Hgb, Platelets, ESR, CRP, Albumin), endoscopic (disease score, pathological activity) and radiological features (bowel wall thickening, enhancement, edema, mesenteric inflammation).

ELIGIBILITY:
Inclusion Criteria:

* Calprotectin assay at IU in last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who had calprotectin assays as part of their evaluations for lower gastrointestinal symptoms in the Division of Gastroenterology at IU within the last 12 months will be considered eligible for the study.
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2006-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chiorean, M.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States